CLINICAL TRIAL: NCT03556124
Title: Imaging-guided tDCS Therapy in Major Depression
Brief Title: Transcranial Direct Current Stimulation in Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Katherine Narr, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-000779; R61MH110526 (NIH)
Record Dates: First submitted 2018-06-02; First posted 2018-06-14 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Major Depressive Disorder
Keywords: Transcranial direct current stimulation; major depression; MRI
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Active and Sham controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active - HD tDCS (Experimental): Participants randomized to this arm will receive 12 sessions of high definition tDCS (HD-tDCS) stimulation (Soterix Medical) delivered to the left dorsolateral prefrontal cortex for 20-30 minutes.
  Interventions: Device: Active - HD tDCS
- Active - Conventional tDCS (Experimental): Participants randomized to this arm will receive 12 sessions of conventional tDCS (C-tDCS) stimulation (Soterix Medical) delivered to the left dorsolateral prefrontal cortex for 20-30 minutes.
  Interventions: Device: Active - Conventional tDCS
- Sham - HD tDCS (Sham Comparator): Participants randomized to this arm will receive 12 sessions of sham HD tDCS stimulation (Soterix Medical) delivered to the left dorsolateral prefrontal cortex for 20-30 minutes.
  Interventions: Device: Sham - HD tDCS
- Sham - Conventional tDCS (Sham Comparator): Participants randomized to this arm will receive 12 sessions of sham conventional tDCS stimulation (Soterix Medical) delivered to the left dorsolateral prefrontal cortex for 20-30 minutes.
  Interventions: Device: Sham - Conventional tDCS

INTERVENTIONS:
Device: Active - HD tDCS — Non-invasive neuromodulation using HD electrodes placed on the scalp to deliver a constant, low current at 2 mA.
  Arms: Active - HD tDCS
Device: Sham - HD tDCS — Sham neuromodulation using HD electrodes placed on the scalp to deliver a low current ramped up/down for 20 sec.
  Arms: Sham - HD tDCS
Device: Active - Conventional tDCS — Non-invasive neuromodulation using standard 7 cm x 5 cm electrodes placed on the scalp to deliver a constant, low current at 2 mA.
  Arms: Active - Conventional tDCS
Device: Sham - Conventional tDCS — Sham neuromodulation using standard 7 cm x 5 cm electrodes electrodes placed on the scalp to deliver a low current ramped up/down for 20 sec.
  Arms: Sham - Conventional tDCS

SUMMARY:
Noninvasive transcranial direct current stimulation (tDCS) is a low-intensity neuromodulation technique of minimal risk that has been used as an experimental procedure for reducing depressive symptoms and symptoms of other brain disorders. Though tDCS applied to prefrontal brain areas is shown to reduce symptoms in some people with major depressive disorder (MDD), the extent of antidepressant response often differs. Methods that map current flow directly in the brain while a person is receiving tDCS and that determine how functional neuroimaging signal changes after a series of tDCS sessions may help us understand how tDCS works, how it can be optimized, and if it can be used as an effective intervention for reducing depressive symptoms. We will investigate these questions in a two-part randomized double blind exploratory clinical trial. The first part of the trial will compare how current flow and functional imaging signal differs in the brain when using tDCS with more focal stimulation, called high definition (HD) tDCS, compared to conventional tDCS (C-tDCS) or sham (non-active) tDCS in patients with MDD.

Sixty people with depression (20 in each group) will be randomized to receive either HD-tDCS, C-tDCS or sham-tDCS for a total of 12 sessions each lasting 20 minutes occurring on consecutive weekdays. At the first and last session, subjects will receive 20-30 minutes of active or sham tDCS in the MRI scanner, which will allow us to map tDCS currents, and track changes in regional cerebral blood flow (rCBF) pre-to- post treatment using completely non-invasive methods. At the first and last session and mid-way through the trial, participants will also complete a series of clinical ratings and neurocognitive tests

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS), a noninvasive neuromodulation technique, applied to the left dorsolateral prefrontal cortex (DLPFC) can reduce depressive symptoms and improve cognitive control in major depressive disorder (MDD). Such findings suggest modulation of top down prefrontal-limbic circuits, which are functionally distinct from ventro-limbic networks and include reciprocally connected DLPFC and dorsomedial anterior cingulate cortex (dACC). However, substantial variation in tDCS response is observed in MDD. This may be due to imprecise stimulation protocols and suboptimal engagement of the neural circuits mediating antidepressant response. Methods that optimize electrode placement and account for individual variation in anatomy and that map current flow directly in the brain may inform the mechanisms and potential clinical utility of tDCS. A new tDCS technique, high definition (HD) tDCS, offers more focal stimulation than conventional tDCS (C-tDCS). The degree to which C-tDCS or HD-tDCS engage dorsal prefrontal-limbic neural circuits is unknown, yet is vital for understanding, confirming and subsequently improving possible therapeutic effects. Innovative MRI techniques that are able to map tDCS currents in vivo and that track changes in regional cerebral blood flow occurring with tDCS over time can provide direct evidence of neural effects. Based on a) theoretical modeling of tDCS current flow, b) studies showing hypo-metabolism, decreased CBF or activity in dorsal prefrontal-limbic networks, c) modulation of these regions with treatment, and, c) our prior results showing significant relationships in between change in dACC rCBF and clinical response to electroconvulsive therapy (ECT), an established brain stimulation treatment, we will test for the tDCS engagement and modulation of the DLPFC and dACC using tDCS current mapping performed in vivo and perfusion MRI. MRI-guided neuronavigation will be used to optimize and standardize electrode placement for DLPFC stimulation.

In this trial we will test for the target engagement of the DLPFC and dACC by comparing C-tDCS, HD-tDCS and sham tDCS applied to the left DLPFC in patients with moderate to severe MDD before and after they complete 12 daily 20-minute sessions of C-tDCS, HD-tDCS or Sham tDCS (n=20 randomized to each group). In-vivo electric current mapping performed at different current intensities (0-2 mA) for 20-30 minutes, and change in regional cerebral blood flow (rCBF) measured before and after a 12-day tDCS trial will determine acute and longer-term modulation of DLPFC and dACC circuitry for each tDCS modality respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 55 years, inclusive
* Gender: all
* Race/ethnicity: all races and ethnic groups
* Capacity to provide informed consent
* Hamilton Rating Scale for Depression (HAMD) score of ≥14 and <24, with or without symptoms of anxiety
* Treatment naïve or on a stable standard antidepressant regimen (including selective serotonin reuptake inhibitors (SSRIs), serotonin-noradrenaline reuptake inhibitors (SNRIs), monoamine oxidase inhibitors (MOAIs) or tricyclic's (TCAs)) with no change in treatment 6-weeks prior to and during the tDCS intervention
* Live within traveling distance to the University of California, Los Angeles (UCLA)

Exclusion Criteria:

* Pregnancy
* Non-English speaking
* Current Substance Use Disorder
* Neurological condition associated with brain abnormalities (e.g., traumatic brain injury; recent stroke, tumor)
* Any contraindication to tDCS (e.g., skin disease or treatment causing irritation)
* Any condition that would contraindicate MRI scanning (metal implants, claustrophobia or a breathing or movement disorder)
* Currently receiving any form of Cognitive Behavioral Therapy, Dialectical Behavioral Therapy, or Acceptance and Commitment Therapy
* Change in antidepressant medication within 6-weeks of starting the trial
* Severe or treatment resistant depression - HAMD scores > 24 and a history of a major depressive episode lasting >2-years or failure to 2 or more antidepressant trials in the current index episode
* Any neuromodulation therapy (e.g., ECT, transcranial magnetic stimulation (rTMS), tDCS) within the last 3-months
* Current or past (within the last 1-month) use of anticonvulsants, lithium, psychostimulant, dexamphetamine
* Current use of decongestants or other medication including sleeping aids previously shown to interfere with cortical excitability
* Schizophrenia Axis I disorder
* Dementia of any type
* Bipolar I disorder
* Diagnosis of seizure disorder or history of seizures
* Depression related to serious medical illness (i.e., mood disorder due to general medical condition)
* Actively suicidal as defined by a score of 4 on item 3 of HAMD

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in non-invasive MRI measures of cerebral blood flow between baseline and end of treatment | Up to 3 weeks
  Modulation of the left dorsolateral prefrontal cortex (DLPFC) and dorsal anterior cingulate cortex (dACC) measured by percent rCBF signal change
Change in non-invasive MRI measures of current flow | 1 hour
  tDCS-induced in vivo magnetic field changes in the left DLPFC as the current is being ramped up from 0 to 2 mA in increments of 0.5 mA over the course of a 1-hour MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Narr, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jog MA, Anderson C, Kubicki A, Boucher M, Leaver A, Hellemann G, Iacoboni M, Woods R, Narr K. Transcranial direct current stimulation (tDCS) in depression induces structural plasticity. Sci Rep. 2023 Feb 17;13(1):2841. doi: 10.1038/s41598-023-29792-6. PMID 36801903
- [Derived] Jog M, Anderson C, Kim E, Garrett A, Kubicki A, Gonzalez S, Jann K, Iacoboni M, Woods R, Wang DJ, Narr KL. A novel technique for accurate electrode placement over cortical targets for transcranial electrical stimulation (tES) clinical trials. J Neural Eng. 2021 Oct 11;18(5):10.1088/1741-2552/ac297d. doi: 10.1088/1741-2552/ac297d. PMID 34555822